CLINICAL TRIAL: NCT04408508
Title: Safety and Efficacy of an Oral Penicillin Challenge in Low Risk Hospitalized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB-19-97
Record Dates: First submitted 2020-02-03; First posted 2020-05-29 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Penicillin Allergy
Keywords: beta-lactam; penicillin; hypersensitivity; drug allergy
MeSH Terms: conditions — Hypersensitivity; Drug Hypersensitivity | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Patients reporting penicillin allergy will be enrolled based on eligibility criteria for direct oral amoxicillin challenge. There will be one treatment group of patients assigned low risk for penicillin allergy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amoxicillin administration (Other): Oral amoxicillin administered to study patients
  Interventions: Drug: Amoxicillin 250 MG

INTERVENTIONS:
Drug: Amoxicillin 250 MG — Low dose oral amoxicillin will be administered to patients enrolled in the study meeting the inclusion and exclusion criteria.
  Other Names: Amoxicillin 250 mg Capsule

SUMMARY:
Penicillin allergy is the most common drug allergy reported by patients. Approximately 10% of the population and 20% of inpatients carry a label of penicillin allergy. However, less than 5%-10% of them have a confirmed allergy following comprehensive investigations. Reported penicillin allergy leads to higher medical costs and excess complications and presents a major challenge to antimicrobial stewardship.

There is a high demand for allergy services however penicillin allergy testing (including skin testing and oral drug challenge) is not routinely available for inpatients even in major centres. Direct oral amoxicillin challenges are safe and effective in delabeling low risk patients who report penicillin allergy in large paediatric and adult studies and does not necessitate specialist referral.

The study team seeks to determine the safety and efficacy of a single-dose oral penicillin challenge pilot program in adult in-patients with self-reported penicillin allergy admitted to hospital under the internal medicine Clinical Teaching Unit (CTU). The study investigators will determine the number of patients successfully delabelled of their "penicillin allergy" prior to discharge from hospital over a 12 month period. The study doctors will also assess the economic impact of the investigator's model and ease of implementation in the busy inpatient setting. In the future this model could be implemented generally as an inpatient or outpatient penicillin allergy program where low risk patients, who do not require referral to an allergist, are expeditiously delabelled.

DETAILED DESCRIPTION:
Penicillin allergy is the most common drug allergy reported by patients. Approximately 10% of the population and 20% of inpatients carry a label of penicillin allergy. However, only <5%-10% of them have a confirmed allergy following comprehensive investigations. Reported penicillin allergy leads to higher medical costs and excess complications and presents a major challenge to antimicrobial stewardship. There is a high demand for allergy services however penicillin allergy testing (including skin testing and oral drug challenge) is not routinely available for inpatients even in major centres. Consequently, patients with a penicillin allergy label receive alternative antibiotics such as carbapenems, fluoroquinolones, and vancomycin for the treatment of common and serious infections and for pre-surgical prophylaxis. Patients with penicillin allergy label have longer hospital stays and higher rates of infections with Clostridioides (Clostridium) difficile, VRE and MRSA in comparison with patients without a documented allergy.

Direct oral amoxicillin challenges are safe and effective in delabeling patients stratified as low risk for penicillin allergy in large pediatric and adult studies. Low-risk penicillin allergy histories include patients who have had isolated nonallergic symptoms (eg, gastrointestinal symptoms) or patients solely with a family history of a penicillin allergy, pruritus without rash, or remote (>10 years) unknown reactions without features suggestive of an IgE-mediated reaction.

The study investigators seek to determine the safety and efficacy of a single-dose oral penicillin challenge pilot program in adult in-patients with self-reported penicillin allergy admitted to hospital under the internal medicine Clinical Teaching Unit (CTU). Identified patients that fulfill the exclusion and inclusion criteria will be reviewed at the time of discharge for suitability, as per the algorithm, modelled after a previous study of similar design. Based on patient's reported allergy, and upon obtaining informed consent, participants will receive a supervised challenge of amoxicillin 250 mg once orally and subsequently observed for 1 hour before discharge home. After antibiotic challenge, patient outcome will be defined as (1) tolerated oral challenge with no adverse drug reaction or (2) adverse drug reaction.

By challenging carefully selected low risk patient that are unlikely to be truly allergic while in hospital, the study doctors can delabel patients of their "penicillin allergy" and as a result cut health care expenditures and promote good antimicrobial stewardship. In the future this model could be implemented generally as an inpatient or outpatient penicillin allergy program where low risk patients, who do not require referral to an allergist, are expeditiously delabeled.

ELIGIBILITY:
Inclusion Criteria:

1. Assessed to be low risk of having a penicillin allergy as per the risk stratification questionnaire
2. One of the following: i) An unknown reaction >10 years before, ii) A type A adverse drug reaction (pharmacologically predictable drug side effect or intolerance), or iii) A history of a benign childhood rash, nonurticarial rash, or maculopapular exanthem more than 10 years ago
3. Age 18 years or older
4. Hemodynamically stable and suitable for discharge home

Exclusion Criteria:

1. Declines participation in the study
2. Cognitive impairment and where a collateral history could not be obtained
3. History of anaphylaxis or angioedema attributed to a penicillin-based antibiotic
4. History of severe cutaneous adverse reactions attributed to a penicillin-based antibiotic
5. History of acute kidney injury or severe liver impairment attributed to a penicillin-based antibiotic
6. Currently taking an angiotensin-converting enzyme inhibitor, angiotensin-receptor blocker or a beta blocker
7. Hemodynamically unstable
8. History of idiopathic urticaria or idiopathic anaphylaxis
9. Currently taking an antibiotic(s) for treatment of an active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients tolerating oral amoxicillin challenge | 12 months
  The number of patients tolerating a single dose oral amoxicillin (250 mg) challenge without adverse reaction(s) up to one hour of administration

SECONDARY OUTCOMES:
Number of patients reporting a delayed reaction to amoxicillin | 12 months
  Number of patients reporting a delayed reaction to amoxicillin (between 1 hour - 12 weeks) following observation and discharge from hospital
Average delay in discharge attributable to amoxicillin challenge | 12 months
  Average delay in discharge (minutes) attributable to penicillin challenge, recorded by the resident or staff physician performing the questionnaire
The number of patients excluded from the study due to staff time constraints | 12 months
  Number of patients excluded from the study due to resident/staff time constraints
Type of immediate reaction attributed to the oral amoxicillin: maculopapular rash, urticaria, angioedema, airway compromise, diarrhea, vomiting or other (including subjective symptoms) | 12 months
  Nature of immediate adverse reaction if challenge unsuccessful

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Fong, MD, FRCPC, Principal Investigator — Saskatchewan Health Authority - Regina Area

IPD SHARING:
Plan to Share IPD: No
No only agregate data will be shared

REFERENCES:
- [Background] Joint Task Force on Practice Parameters; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. Drug allergy: an updated practice parameter. Ann Allergy Asthma Immunol. 2010 Oct;105(4):259-273. doi: 10.1016/j.anai.2010.08.002. PMID 20934625
- [Result] Macy E. Penicillin allergy: optimizing diagnostic protocols, public health implications, and future research needs. Curr Opin Allergy Clin Immunol. 2015 Aug;15(4):308-13. doi: 10.1097/ACI.0000000000000173. PMID 26110680
- [Result] Macy E, Ngor EW. Safely diagnosing clinically significant penicillin allergy using only penicilloyl-poly-lysine, penicillin, and oral amoxicillin. J Allergy Clin Immunol Pract. 2013 May-Jun;1(3):258-63. doi: 10.1016/j.jaip.2013.02.002. Epub 2013 Apr 6. PMID 24565482
- [Result] Mohamed OE, Beck S, Huissoon A, Melchior C, Heslegrave J, Baretto R, Ekbote A, Krishna MT. A Retrospective Critical Analysis and Risk Stratification of Penicillin Allergy Delabeling in a UK Specialist Regional Allergy Service. J Allergy Clin Immunol Pract. 2019 Jan;7(1):251-258. doi: 10.1016/j.jaip.2018.05.025. Epub 2018 Jun 5. PMID 29883754
- [Result] Macy E, Contreras R. Health care use and serious infection prevalence associated with penicillin "allergy" in hospitalized patients: A cohort study. J Allergy Clin Immunol. 2014 Mar;133(3):790-6. doi: 10.1016/j.jaci.2013.09.021. Epub 2013 Nov 1. PMID 24188976
- [Result] Mill C, Primeau MN, Medoff E, Lejtenyi C, O'Keefe A, Netchiporouk E, Dery A, Ben-Shoshan M. Assessing the Diagnostic Properties of a Graded Oral Provocation Challenge for the Diagnosis of Immediate and Nonimmediate Reactions to Amoxicillin in Children. JAMA Pediatr. 2016 Jun 6;170(6):e160033. doi: 10.1001/jamapediatrics.2016.0033. Epub 2016 Jun 6. PMID 27043788
- [Result] Tucker MH, Lomas CM, Ramchandar N, Waldram JD. Amoxicillin challenge without penicillin skin testing in evaluation of penicillin allergy in a cohort of Marine recruits. J Allergy Clin Immunol Pract. 2017 May-Jun;5(3):813-815. doi: 10.1016/j.jaip.2017.01.023. Epub 2017 Mar 21. No abstract available. PMID 28341170
- [Result] Labrosse R, Paradis L, Lacombe-Barrios J, Samaan K, Graham F, Paradis J, Begin P, Des Roches A. Efficacy and Safety of 5-Day Challenge for the Evaluation of Nonsevere Amoxicillin Allergy in Children. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1673-1680. doi: 10.1016/j.jaip.2018.01.030. Epub 2018 Feb 7. PMID 29425903
- [Result] Iammatteo M, Alvarez Arango S, Ferastraoaru D, Akbar N, Lee AY, Cohen HW, Jerschow E. Safety and Outcomes of Oral Graded Challenges to Amoxicillin without Prior Skin Testing. J Allergy Clin Immunol Pract. 2019 Jan;7(1):236-243. doi: 10.1016/j.jaip.2018.05.008. Epub 2018 May 23. PMID 29802906
- [Result] Ibanez MD, Rodriguez Del Rio P, Lasa EM, Joral A, Ruiz-Hornillos J, Munoz C, Gomez Traseira C, Escudero C, Olaguibel Rivera JM, Garriga-Baraut T, Gonzalez-de-Olano D, Rosado A, Sanchez-Garcia S, Perez Bustamante S, Padial Vilchez MA, Prieto Montano P, Candon Morillo R, Macias Iglesia E, Feliu Vila A, Valbuena T, Lopez-Patino A, Martorell A, Sastre J, Audicana MT; Penicillin Allergy in Children (APENIN) Task Force. Pediatric Allergy Committee, Spanish Society of Allergy and Clinical Immunology (SEAIC). Prospective assessment of diagnostic tests for pediatric penicillin allergy: From clinical history to challenge tests. Ann Allergy Asthma Immunol. 2018 Aug;121(2):235-244.e3. doi: 10.1016/j.anai.2018.05.013. Epub 2018 May 25. PMID 29803713
- [Result] Confino-Cohen R, Rosman Y, Meir-Shafrir K, Stauber T, Lachover-Roth I, Hershko A, Goldberg A. Oral Challenge without Skin Testing Safely Excludes Clinically Significant Delayed-Onset Penicillin Hypersensitivity. J Allergy Clin Immunol Pract. 2017 May-Jun;5(3):669-675. doi: 10.1016/j.jaip.2017.02.023. PMID 28483317
- [Result] Banks TA, Tucker M, Macy E. Evaluating Penicillin Allergies Without Skin Testing. Curr Allergy Asthma Rep. 2019 Mar 22;19(5):27. doi: 10.1007/s11882-019-0854-6. PMID 30903298